CLINICAL TRIAL: NCT05001126
Title: The Effects of High Intensity Functional Training on Cardiometabolic Risk Factors and Exercise Enjoyment in Men and Women With Metabolic Syndrome: a Randomized, 12-week, Dose-response Trial
Brief Title: The Dose-response Effects of High Intensity Functional Training on Metabolic Syndrome Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary Van Guilder (Other)
Collaborators: Western Colorado University (Other); Auckland University of Technology (Other)
Responsible Party: Sponsor-Investigator, Gary Van Guilder, Sponsor Investigator, Western Colorado University
Organization: Western Colorado University (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: WCU_HIFT_MetS
Record Dates: First submitted 2021-07-14; First posted 2021-08-11 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Metabolic Syndrome; Atherogenic Dyslipidemia; Insulin Resistance; Endothelial Dysfunction
Keywords: Exercise
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Motor Activity

STUDY DESIGN:
Intervention Model Description: Three dose groups
Who Masked: Investigator
Masking Description: Primary investigator will be blinded from each participant's dose allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIFT 1x/week (Experimental): HIFT exercise performed one time per week.
  Interventions: Behavioral: HIFT 1x/week
- HIFT 2x/week (Experimental): HIFT exercise performed two times per week.
  Interventions: Behavioral: HIFT 2x/week
- HIFT 3x/week (Experimental): HIFT exercise performed three times per week.
  Interventions: Behavioral: HIFT 3x/week

INTERVENTIONS:
Behavioral: HIFT 1x/week — HIFT is a time-efficient modality of exercise combining high-intensity aerobic and resistance training using minimal equipment. HIFT 1x/week represents a dose of one HIFT workout per week.
  Arms: HIFT 1x/week
Behavioral: HIFT 2x/week — HIFT is a time-efficient modality of exercise combining high-intensity aerobic and resistance training using minimal equipment. HIFT 2x/week represents a dose of two HIFT workouts per week.
  Arms: HIFT 2x/week
Behavioral: HIFT 3x/week — HIFT is a time-efficient modality of exercise combining high-intensity aerobic and resistance training using minimal equipment. HIFT 3x/week represents a dose of three HIFT workouts per week.
  Arms: HIFT 3x/week

SUMMARY:
This study aims to explore the dose effects of three weekly volumes of high-intensity functional training (HIFT) on apolipoprotein B (ApoB), triglyceride (TG) and cholesterol (CHOL) content of low-density lipoproteins (LDL), very low-density lipoproteins (VLDL), and high-density lipoproteins (HDL) particles, fasting insulin and glucose, glycosylated hemoglobin (HbA1c), and endothelial function after a 12-week training program. Secondarily, this study aims to also explore the subjective dose-responses of "exercise enjoyment" and "intention to continue" after this 12-week training program.

DETAILED DESCRIPTION:
Background: Individuals with metabolic syndrome (MetS) are at a greater risk for developing atherosclerotic cardiovascular disease (ASCVD) than those without MetS, due to underlying endothelial dysfunction, dyslipidemia, and insulin resistance. Exercise is an effective primary and secondary prevention strategy for MetS, however less than 25% of adults meet the minimum stated public recommendations. Barriers often identified are lack of enjoyment and lack of time. High intensity functional training (HIFT), a time efficient modality of exercise, has shown some potential to elicit positive affectivity, and elicit increased fitness and improved glucose metabolism. However, the effects of HIFT on dyslipidemia and endothelial dysfunction have not been explored, nor have the effects been explored in a population with MetS. Additionally, no studies have investigated the minimal dose of HIFT per week to see clinically meaningful changes in cardiometabolic health. The purpose of this study is to: 1) determine the dose-response effect of HIFT on blood lipids, insulin resistance, and endothelial function, and 2) determine the dose-response effect of HIFT on body composition, fitness, and perceived enjoyment and intention to continue the exercise.

Methods/design: In this randomized, dose-response trial, participants will undergo a 12-week HIFT intervention of either 1 day/week, 2 days/week, or 3 days/week of supervised, progressive exercise. Outcomes assessed at baseline and post-intervention will be multiple cardiometabolic markers, and fitness. Additionally, the participant's affective response will be measured after the intervention.

Discussion: The findings of this research will provide evidence on the minimal dose of HIFT per week to see clinically meaningful improvements in the risk factors of MetS, as well as whether this modality is likely to mitigate the barriers to exercise. If an effective dose of HIFT per week is determined and if this modality is perceived positively, it may provide exercise specialists and health care providers a tool to prevent and treat MetS.

ELIGIBILITY:
Inclusion Criteria:

* Physically Inactive (< 30 min/day, 3 days/wk, for 3 months of moderate intensity exercise)
* Possess at least 3 of the following 5 risk factors defining metabolic syndrome (MetS): waist circumference ≥ 102cm (men) or ≥ 88cm (women), resting blood pressure ≥ 130/85, HDL-C ≤ 40mg/dl (men) or ≤ 50mg/dl (women), fasting triglycerides ≥ 150mg/dl, and fasting blood glucose ≥ 100mg/dl.

Exclusion Criteria:

* Diagnosed heart, lung, kidney, liver, pancreatic or neurological disease
* Pregnant or plan to become pregnant
* Medical or orthopedic conditions preventing participation in exercise

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline and comparison between groups in apolipoprotein B (ApoB) count after 12 weeks of training. | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of apolipoprotein B will be measured via venipuncture of the anti-cubital vein and reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in the cholesterol content of low-density lipoproteins (LDL-C). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of LDL-C will be measured via venipuncture of the anti-cubital vein and reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in the cholesterol content of very low-density lipoproteins (VLDL-C). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of VLDL-C will be measured via venipuncture of the anti-cubital vein and reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in the cholesterol content of high-density lipoproteins (HDL-C). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of HDL-C will be measured via venipuncture of the anti-cubital vein and reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in the total cholesterol (TC) content of all lipoproteins. | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of TC will be measured via venipuncture of the anti-cubital vein and reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in the triglyceride content of LDL (LDL-T). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of LDL-T will be measured via venipuncture of the anti-cubital vein and reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in the triglyceride content of VLDL (VLDL-T). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of VLDL-T will be measured via venipuncture of the anti-cubital vein and reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in the total triglyceride content of all lipoprotein classes (TG). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of TG will be measured via venipuncture of the anti-cubital vein and reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in blood glucose (BG). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of BG will be measured via venipuncture of the anti-cubital vein and reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change for each variable will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in blood insulin (INS). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of INS will be measured via venipuncture of the anti-cubital vein and reported in units of mcIU/mL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change for each variable will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in the Homeostatic Assessment of Insulin Resistance (HOMA-IR). | Baseline and 48hrs post 12-week training completion
  The baseline and post-training blood analysis of BG and INS will be used to calculate insulin resistance (IR) using the validated homeostatic model assessment (HOMA) [Sarafidis et al., 2007; Matthews et al., 1985]. HOMA-IR will be reported in units of mg/dL. Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change for each variable will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in glycosylated hemoglobin (HbA1c) after 12 weeks of training. | Baseline and 48hrs post 12-week training completion
  Baseline and post-training blood analysis of HbA1c will be measured via venipuncture of the anti-cubital vein and reported in units of percent (%). Change from baseline will be calculated and aggregated as mean (SD) for each dose group as well as for male and female subgroups within each dose group. The mean (SD) change for each variable will be compared between the three dose groups and male and female subgroups.
Mean change from baseline and comparison between groups of endothelial-dependent peak blood flow (PBF). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training endothelial-dependent PBF of the non-dominant forearm will be measured using venous occlusion strain-gauge plethysmography and reported in units of percent (%). Change from baseline will be calculated and aggregated as mean (SD) for each dose group and male/female subgroups. Mean (SD) for each variable will be compared between dose groups and male and female subgroups.
Mean change from baseline and comparison between groups of endothelial-dependent area under the curve (AUC) of hyperemia blood flow. | Baseline and 48hrs post 12-week training completion
  Baseline and post-training endothelial-dependent hyperemia AUC of the non-dominant forearm will be measured using venous occlusion strain-gauge plethysmography. Hyperemia blood flow will be measured for 5 min after a 5 min occlusion period. 30 sec AUC blood flow will be quantified reported in units of percent (%) x time. Change from baseline will be calculated and aggregated as mean (SD) for each dose group and male/female subgroups. Mean (SD) for each variable will be compared between dose groups and male and female subgroups.

SECONDARY OUTCOMES:
Mean change from baseline and comparison between groups of body fat mass percentage (FM%). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training FM% will be measured via dual X-ray absorptiometry (DEXA) and reported as percentage of total body mass. Change from baseline will be calculated and aggregated as mean (SD) for each dose group and male and female subgroups. Mean (SD) will be compared between dose groups and male and female subgroups.
Mean change from baseline and comparison between groups of body lean mass percentage (LM%). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training LM% will be measured via dual X-ray absorptiometry (DEXA) and reported as percentage of total body mass. Change from baseline will be calculated and aggregated as mean (SD) for each dose group and male and female subgroups. Mean (SD) will be compared between dose groups and male and female subgroups.
Mean change from baseline and comparison between groups in maximal oxygen consumption (VO2max). | Baseline and 48hrs post 12-week training completion
  Baseline and post-training VO2max will be measured via a graded exercise test (GXT) on a power treadmill. After a 5 min warm-up, participants will walk at a constant speed while incline is increased 1% each minute until volitional exhaustion [Balke & Ware, 1959] while VO2 is continuously captured. VO2max will be recorded and reported in units of mL/kg/min. Participants will rest passively for 20 min then perform a verification trial at 105% of their maximal GXT workload while VO2 is continuously captured until volitional exhaustion. If VO2max of the verification bout and GXT are within ± 3%, true VO2max will be considered achieved [Astorino et al., 2009; Nolan et al., 2014; Weatherwax et al., 2016]. If verification is not achieved, they will repeat the trial after a 24hr rest. Change from baseline will be calculated and aggregated as mean (SD) for each dose group and male/female subgroups. Mean (SD) will be compared between the three dose groups and male/female subgroups.
Mean change from baseline and comparison between groups of self-perceived fitness after 12 weeks of training. | Baseline and 48hrs post 12-week training completion
  Baseline and post-training self-perceived fitness will be measured using the validated International Fitness Scale (IFIS) [Ortega et al., 2011; Merellano-Navarro et al., 2017] and reported as the sum of all scores. The scale contains five questions with the answering options (Very Poor-1, Poor-2, Average-3, Good-4, Very Good-5) associated to these elements of physical fitness: cardiorespiratory endurance, muscular strength, speed-agility, and flexibility. Change from baseline will be calculated and aggregated as mean (SD) for each dose group and male/female subgroups. Mean (SD) will be compared between the three dose groups and male/female subgroups.

OTHER OUTCOMES:
Comparison between groups of exercise enjoyment perception after 12 weeks of training. | 24hrs post 12-week training completion
  To assess the participants perception of enjoyment of their allocated HIFT intervention, the validated Physical Activity Enjoyment Scale (PACES) will be used [Kendzierski & DeCarlo, 1991] and reported as the sum of all scores. The PACES is an 18-item, 7-point bipolar rating scale where 1 represents the lowest level of enjoyment and 7 represents the highest level of enjoyment. Data will be aggregated as mean (SD) for each dose group and male/female subgroups. Mean (SD) will be compared between dose groups and male/female subgroups.
Comparison between groups of the intention to continue their allocated intervention after 12 weeks of training. | 24hrs post 12-week training completion
  To assess the participants intention to continue their allocated HIFT intervention, two additional items will be added to the PACES regarding 1) how likely the participant will continue performing the modality of exercise (0=unlikely to 10=very likely) and 2) how many days per week the participant will would consider performing the modality of exercise (0-7 days) [Kwan & Bryan, 2010; Heinrich et al., 2019]. Data per question will be aggregated as mean (SD) for each dose group and male/female subgroups. Mean (SD) will be compared between dose groups and male/female subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Lance C Dalleck, PhD, Principal Investigator — Western Colorado University; Nigel Harris, PhD, Principal Investigator — Auckland University of Technology
Locations (1):
- Western Colorado University, Gunnison, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available upon request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available indefinitely upon completion of trail and statistical analysis.
Access Criteria: Data will be available upon request via email to principle investigator.

REFERENCES:
- [Background] Sarafidis PA, Lasaridis AN, Nilsson PM, Pikilidou MI, Stafilas PC, Kanaki A, Kazakos K, Yovos J, Bakris GL. Validity and reproducibility of HOMA-IR, 1/HOMA-IR, QUICKI and McAuley's indices in patients with hypertension and type II diabetes. J Hum Hypertens. 2007 Sep;21(9):709-16. doi: 10.1038/sj.jhh.1002201. Epub 2007 Apr 19. PMID 17443211
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Ortega FB, Ruiz JR, Espana-Romero V, Vicente-Rodriguez G, Martinez-Gomez D, Manios Y, Beghin L, Molnar D, Widhalm K, Moreno LA, Sjostrom M, Castillo MJ; HELENA study group. The International Fitness Scale (IFIS): usefulness of self-reported fitness in youth. Int J Epidemiol. 2011 Jun;40(3):701-11. doi: 10.1093/ije/dyr039. Epub 2011 Mar 24. PMID 21441238
- [Background] Merellano-Navarro E, Collado-Mateo D, Garcia-Rubio J, Gusi N, Olivares PR. Validity of the International Fitness Scale "IFIS" in older adults. Exp Gerontol. 2017 Sep;95:77-81. doi: 10.1016/j.exger.2017.05.001. Epub 2017 May 2. PMID 28476584
- [Background] BALKE B, WARE RW. The present status of physical fitness in the Air Force. Proj Rep USAF Sch Aviat Med. 1959 May;59(67):1-9. No abstract available. PMID 24546008
- [Background] Astorino TA, White AC, Dalleck LC. Supramaximal testing to confirm attainment of VO2max in sedentary men and women. Int J Sports Med. 2009 Apr;30(4):279-84. doi: 10.1055/s-0028-1104588. Epub 2009 Feb 6. PMID 19199208
- [Background] Nolan PB, Beaven ML, Dalleck L. Comparison of intensities and rest periods for VO2max verification testing procedures. Int J Sports Med. 2014 Nov;35(12):1024-9. doi: 10.1055/s-0034-1367065. Epub 2014 Jun 2. PMID 24886925
- [Background] Weatherwax RM, Richardson TB, Beltz NM, Nolan PB, Dalleck L. Verification Testing to Confirm VO2max in Altitude-Residing, Endurance-Trained Runners. Int J Sports Med. 2016 Jun;37(7):525-30. doi: 10.1055/s-0035-1569346. Epub 2016 Apr 29. PMID 27128112
- [Background] Kendzierski D and DeCarlo KJ. Physical activity enjoyment scale: Two validation studies. Journal of Sport and Exercise Psychology. 1991; 13:50-64.
- [Background] Kwan BM, Bryan A. In-task and post-task affective response to exercise: translating exercise intentions into behaviour. Br J Health Psychol. 2010 Feb;15(Pt 1):115-31. doi: 10.1348/135910709X433267. Epub 2009 Apr 25. PMID 19397847
- [Background] Heinrich KM, Crawford DA, Johns BR, Frye J, and Gilmore KEO. Affective responses during high-intensity functional training compared to high-intensity interval training and moderate continuous training. Sport, Exercise, and Performance Psychology. 2019;9(1):115-127.
- [Derived] Smith LE, Van Guilder GP, Dalleck LC, Harris NK. The effects of high-intensity functional training on cardiometabolic risk factors and exercise enjoyment in men and women with metabolic syndrome: study protocol for a randomized, 12-week, dose-response trial. Trials. 2022 Mar 1;23(1):182. doi: 10.1186/s13063-022-06100-7. PMID 35232475